CLINICAL TRIAL: NCT07105540
Title: Comparison of Hydrodissection With 5% Dextrose and Perineural Corticosteroid Injection in Carpal Tunnel Syndrome: A Prospective Study
Brief Title: Comparison of Injection Techniques in Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Gizem Suna Tuncer, Principal Investigator, Physical Medicine and Rehabilitation Specialist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AE-FTR-GST-01
Record Dates: First submitted 2025-07-14; First posted 2025-08-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Hydrodissection; Perineural Injection; Median Nerve
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Glucose; Betamethasone; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrodissection group (Active Comparator): Participants in the hydrodissection group will undergo ultrasound-guided perineural hydrodissection of the median nerve at the scaphoid-pisiform level using a 12 MHz linear transducer (GE Logiq P9, GE Healthcare, Boston, MA). Under sterile conditions, 2.5 ml of 5% dextrose will be injected via an in-plane ulnar approach to mechanically separate the median nerve from the transverse carpal ligament. Subsequently, an additional 2.5 ml of 5% dextrose will be administered to separate the nerve from adjacent flexor tendons. The total injection volume will be 5 ml.
  Interventions: Drug: 5% Dextrose
- Corticosteroid group (Active Comparator): Participants in the corticosteroid group will undergo ultrasound-guided perineural injection of the median nerve at the scaphoid-pisiform level using a 12 MHz linear transducer (GE Logiq P9, GE Healthcare, Boston, MA). A perineural injection of 1 ml betamethasone combined with 1 ml 2% lidocaine will be administered around the median nerve.
  Interventions: Drug: Betamethasone and local anesthetic

INTERVENTIONS:
Drug: 5% Dextrose — Ultrasound-guided hydrodissection is performed using a 12 MHz linear transducer (GE Logiq P9, GE Healthcare) via an in-plane ulnar approach under sterile conditions. 2.5 ml of 5% dextrose will be injected via an in-plane ulnar approach to mechanically separate the median nerve from the transverse carpal ligament. Subsequently, an additional 2.5 ml of 5% dextrose will be administered to separate the nerve from adjacent flexor tendons. The total injection volume will be 5 ml.
  Arms: Hydrodissection group
Drug: Betamethasone and local anesthetic — Ultrasound-guided perineural injection is performed using a 12 MHz linear transducer (GE Logiq P9, GE Healthcare) via an in-plane ulnar approach under sterile conditions. A total of 2 ml solution (1 ml betamethasone and 1 ml 2% lidocaine) is injected perineurally around the median nerve under ultrasound guidance at the scaphoid-pisiform level.
  Arms: Corticosteroid group

SUMMARY:
The aim of this study is to compare the effects of ultrasound-guided hydrodissection with 5% dextrose and perineural corticosteroid injection on the clinical parameters of carpal tunnel syndrome, as well as to evaluate the long-term efficacy of these treatments.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS), the most prevalent peripheral compressive neuropathy, manifests primarily with sensory disturbances such as pain, numbness, and nocturnal paresthesia. Treatment options for CTS differ considerably depending on the severity of symptoms, and typically include splinting, physiotherapy, local injection therapies, and surgical release. Hydrodissection is an ultrasound-guided technique that has recently gained increased attention for its role in the management of nerve entrapment syndromes. The technique uses fluid injection to separate the nerve from nearby tissues. This may reduce perineural adhesions and improve the patient's symptoms. In hydrodissection, normal saline, 5% dextrose, or platelet-rich plasma (PRP) can be used as injectates. Recently, hydrodissection with 5% dextrose has become the most commonly used approach. Several studies in the literature have demonstrated that perineural hydrodissection with 5% dextrose provides more favorable outcomes than corticosteroid injections in patients with mild to moderate CTS, particularly at 4 to 6 months post-injection. However, it remains unclear whether hydrodissection leads to a reduction in the cross-sectional area of the median nerve. In addition, studies examining the procedural details of hydrodissection are limited. Therefore, further clinical research is needed to better understand and validate the technique.

Ultrasound-guided hydrodissection for CTS is performed using a 12 MHz linear array transducer probe (GE Logiq P9, GE Healthcare, Boston, MA). The median nerve (MN) is visualized at the scaphoid-pisiform level. In the intervention group, 2.5 ml of 5% dextrose is injected via an in-plane ulnar approach to separate the MN from the transverse carpal ligament, followed by an additional 2.5 ml of normal saline (NS) injected to separate the MN from the flexor tendons. In the control group, perineural injection of 1 ml betamethasone is administered around the MN using the same ultrasound device and probe.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with unilateral moderate carpal tunnel syndrome (CTS) confirmed by an electrophysiological study within the last 6 months
* Presence of at least one of the following symptoms lasting more than one month:

  * Paresthesia/dysesthesia accompanied by weakness and clumsiness in the hand, worsened by repetitive wrist use or sleep, and relieved by postural correction or shaking of the hand
  * Numbness due to sensory disturbance in the median nerve (MN) distribution
  * Thenar muscle weakness with atrophy
  * Positive Tinel's sign or Phalen's test
* Pain intensity of ≥4 out of 10 on the Visual Analog Scale (VAS) prior to treatment

Exclusion Criteria:

* History of previous wrist surgery, polyneuropathy, brachial plexopathy, or thoracic outlet syndrome
* Presence of systemic infection
* Pregnancy
* Prior corticosteroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-02-05 (Actual); Study Completion 2026-02-05 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire | At baseline, at Month 1,3,6 (Visit 1,2,3)
  The Boston Carpal Tunnel Questionnaire (BCTQ) is a validated disease-specific assessment tool developed in 1993 to provide standardized clinical evaluation of carpal tunnel syndrome (CTS). It comprises 19 items divided into two subscales: the Symptom Severity Scale (BCTQ-SSS) and the Functional Status Scale (BCTQ-FSS). Scores on both subscales range from 1 to 5, with higher scores reflecting increased symptom burden and functional impairment associated with CTS.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | At baseline and at Month 1,3,6 (Visit 1,2,3)
  Patients rate their pain on a 0-10 scale. A lower score indicates reduced pain.
Cross-Sectional Area (CSA) of the Median Nerve via Ultrasonography | At baseline and at month 3,6 (Visit 2,3)
  Median nerve CSA will be measured at the scaphoid-pisiform level. A reduction in CSA indicates improvement.
Hand Grip Strength | At baseline and at Month 3,6 (Visit 2,3)
  Hand grip strength will be measured using a standard Jamar dynamometer. During the procedure, patients will be seated with the elbow flexed at 90° and the forearm in a neutral position. Three consecutive measurements will be taken, and the average value will be recorded. Improvement reflects functional recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No